CLINICAL TRIAL: NCT05252468
Title: COVID-19 Prevention Trial: Effect of Prophylactic Use of TAFFIX™ on Infection Rate by SARS-CoV-2 Virus (COVID-19).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nasus Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NP-003-Taffix
Record Dates: First submitted 2022-02-10; First posted 2022-02-23 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Upper Respiratory Tract Infections
Keywords: Upper respiratory tract infection; viruses; COVID-19; nasal; powder; prevention; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TaffiX™ (Experimental): TaffiX™ is a Nasal powder personal spray that blocks viruses particles from entering the nasal cells.
  Interventions: Device: TaffiX™
- Lactose powder (Placebo Comparator): Lactose nasal powder will be used as a placebo. It has an identical appearance as TaffiX™ (white powder in an identical bottle).
  Interventions: Device: TaffiX™

INTERVENTIONS:
Device: TaffiX™ — Personal nasal powder spray.

SUMMARY:
TAFFIX is a nasal powder spray that immediately creates a protective acidic barrier on the nasal mucosa against infection by inhaled viruses. The protective barrier lasts 5 hours.

TAFFIX is approved as a medical device in Israel, intended for use to block inhaled viruses within the nasal cavity. In Europe, it is registered as a medical device indicated for use as a protective mechanical barrier against allergens and viruses (e.g., SARS-CoV-2) within the nasal cavity.

TAFFIX is used as additional safety mean together with masks, hygiene, and social distancing.

The study rationale is to evaluate whether daily use of TaffiX™ as prophylaxis will reduce the rate of SARS- CoV-2 infection and other upper respiratory infections, compared to the placebo control rate.

DETAILED DESCRIPTION:
Study Design:

This is a 2 arms, Randomized, double blind, placebo controlled clinical trial.

Study population:

Subjects who, were not diagnosed with COVID-19 previously to their best knowledge and according to COVID-19 antibody test.

Were not vaccinated yet against COVID-19 and will not be vaccinated during their participating in the study.

Up to 1000(500 per study arm) will be enrolled for the purpose of this study.

Study treatment:

TaffiX™ will be used daily (up to 3 times a day, every 5 hours) in addition to the protective measures instructed by the Ministry of Health The control group will be administrated with Placebo- lactose powder for nasal application

Participation duration:

Up to 6 weeks

Concomitant therpay:

Allowed- no restriction for Concomitant Medications

Planned interim analyses:

When no less than 150 subjects have completed the study, an interim analysis for Efficacy and safety will be conducted by an independent biostatistician.

After no less than 500 subjects, additional interim analysis for Efficacy and safety will be conducted by an independent biostatistician.

Serious adverse events will be monitored by an independent safety officer on an ongoing basis throughout the study.

Stop Rule:

If the proportion of COVID-19 positive rate in the treatment group is statistically significantly lower than the proportion of COVID-19 positive rate in the placebo control group.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 12 yr and older who had not previously been infected with COVID-19 to the best of their knowledge.
2. Were not vaccinated yet against COVID-19 and will not be vaccinated during the study (if they decide to get the vaccine during the study they will be excluded a week later).
3. Negative serology rapid test to COVID-19.
4. Be informed of the nature of the study and the procedures and sign an informed consent form.
5. Willing and able to adhere to Protocol requirements.
6. If female of childbearing potential, agree to use an acceptable method of birth control or be surgically sterile, and have a negative pregnancy test.

Exclusion Criteria:

1. Known sensitivity to citric acid and/or sodium citrate and /or benzalkonium chloride and /or Hydroxypropylmethylcellulose (HPMC) or lactose (does not mean diagnosed lactose intolerance in food).
2. Females who are pregnant or are lactating as reported by the subject.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
COVID-19 new cases | Through study completion, 6 weeks
  symptoms score (Fever; Cough; Rigors; Myalgia; Headache; Vomiting or Diarrhea; Shortness of breath; Breathing difficulties; New olfactory and taste disorder(s); Runny or stuffy nose; Sore throat) as reported in Bi-weekly questionnaires, PCR or antigen test at symptomatic subjects, serology test at end of the study.

SECONDARY OUTCOMES:
The safety and tolerability of the study device. | Through study completion, 6 weeks.
  Incidence of adverse events as reported by subjects

OTHER OUTCOMES:
To evaluate the efficacy of Taffix in preventing upper respiratory infection | Through study completion, 6 weeks
  Incidence of symptoms (Fever; Cough; Rigors; Myalgia; Headache; Vomiting or Diarrhea; Shortness of breath; Breathing difficulties; New olfactory and taste disorder(s); Runny or stuffy nose; Sore throat), as reported in Bi-weekly questionnaires, at subjects who were negative to SARS-CoV-2
Severity of COVID-19 | Through study completion, 6 weeks
  Severity of COVID-19 cases (according to NIH severity categories)
Change in Allergic Rhinitis or Asthma symptoms in relevant subjects | Through study completion, 6 weeks
  By report to the study coordinator, among subjects who reported of that condition at the entry to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Emil Kolev, MD, Principal Investigator — Nasus Pharma
Locations (1):
- Diagnostics and Consultation Center Convex Ltd, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No